CLINICAL TRIAL: NCT01064388
Title: A Phase I, Single Center, Double-blind Randomized, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics of Intravenous AZD9742 After Administration of Multiple Ascending Doses for 14 Days in Healthy Male and Female Subjects
Brief Title: A Study in Healthy Volunteers to Assess Safety and Blood Levels of AZD9742 After Multiple Doses Over 14 Days
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2690C00002
Record Dates: First submitted 2010-02-03; First posted 2010-02-08 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Healthy
Keywords: Safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD9742
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD9742 — IV infusion, 15 days
  Arms: 1
Drug: Placebo — IV infusion, 15 days
  Arms: 2

SUMMARY:
The purpose of this study is to determine the safety, tolerability and blood levels of AZD9742 after daily dosing for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 19-30

Exclusion Criteria:

* Positive Fecal Occult Blood Test
* Prescriptions that inhibit liver function
* Received flu/H1N1 vaccine within 2 weeks before first dose

Ages: 23 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Safety variables (adverse events, vital signs, physical examinations, clinical laboratory assessments, 12-lead ECG, digital ECG, telemetry) | collected prior to treatment, during treatment and follow-up for a total of 25-30 days.

SECONDARY OUTCOMES:
To characterize the Pharmacokinetics of AZD9742 in blood and urine | PK-sampling during 14 pre-defined study days for PK profiling

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Shaw, Study Director — AstraZeneca; Brendan Smyth, Study Chair — AstraZeneca; David Melnick, Study Director — AstraZeneca; Ralph Schutz, Principal Investigator — Quintiles, Inc.
Locations (1):
- Research Site, Overland Park, Kansas, United States